CLINICAL TRIAL: NCT07385118
Title: Daily Fluctuations in Brain-Derived Neurotrophic Factor and Cognitive Performance: Effects of Acute Physical Exercise
Brief Title: Daily Fluctuations in Brain-Derived Neurotrophic Factor and Cognition: Effects of Vigorous Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DAILYBDNF
Record Dates: First submitted 2026-01-07; First posted 2026-02-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: BDNF
Keywords: BDNF; Cognition; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BDNF arm (Experimental): Every subject will be tested on day 1 and day 2 with the same protocol. Blood samples will be collected at five time points throughout the workday: 09:00 (T1), 11:00 (T2), 13:00 (T3), 15:00 (T4), and 17:00 (T5), to assess potential diurnal variations in BDNF. Cognitive performance will be evaluated using the Psychomotor Vigilance Test (PVT), the Flanker task, and the Digit Span Backwards test at T1, T3, and T5. On the second intervention day, the same protocol will be followed, with the addition of a 15-minute single bout of high-intensity physical activity executed at T4.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A five-minute bout of exercise at high intensity (75% of HRmax) repeated for two rounds with a minute rest between rounds. The bout consists of 5 exercises: BW squat, jumping jacks, lunges, crunches and step up. The modality is, in one minute for every exercise, 30 seconds of work and 30 seconds of rest

SUMMARY:
Cognitive functions are fundamental to everyday life, underpinning the mental processes required to perform any activity. Recent studies have shown that improved cognitive performance is associated with elevated levels of brain-derived neurotrophic factor (BDNF), which can be increased through an acute bout of physical activity. However, daily variations of BDNF serum and plasma remain poorly characterised and are not fully understood, and their correlation with daily variations in cognitive performance has not been previously explored. This study examines:

1) the correlation between daily BDNF fluctuations and cognitive performance. 2) whether a single session of exercise can elevate BDNF levels and lead to measurable cognitive improvements.

ELIGIBILITY:
Inclusion Criteria:

* an age between 18-40 years old
* no history of mental or physical diseases (of a neurological, psychogenic, musculoskeletal, cardiorespiratory or systemic nature)
* MoCA score higher than 26

Exclusion Criteria:

* smokers
* individuals experiencing sleep-wake cycle disturbances in the week prior to the study
* consumers of medications with CNS effects

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Levels of Serum BDNF (ng/ml) | blood samples were collected on day one and day two at five specific time points: 9 a.m. (t1), 11 a.m. (t2), 1 p.m. (t3), 3 p.m. (t4), 5 p.m. (t5)
  Blood samples for serum BDNF concentration analysis were collected using a Clot Activator Tube (CAT) and gently swirled ten times, upside down. They were then incubated at room temperature for 30 minutes to allow clot formation. Subsequently, the samples were centrifuged at 1100 g and 4 °C for 10 minutes, and then, the serum was collected, aliquoted, and stored at -80 °C. The analysis of BDNF was performed using an enzyme-linked immunosorbent assay (ELISA) kit, following the manufacturer's instructions (ab212166 - Human BDNF SimpleStep ELISA Kit).
inhibitory control | The test was performed for each participant on day one and two at three predefined time points 9 a.m. (t1), 1 p.m. (t3), 5 p.m. (t5)
  Inhibitory control was assessed with the Flanker Task. During the task, participants are required to indicate the left-right orientation of a centrally presented stimulus while inhibiting attention to the potentially incongruent stimuli surrounding it (e.g., flankers on either side). The principal outcomes for this task are total errors, the mean reaction time for incongruent and congruent stimuli, and the conflict cost (the difference between the mean reaction times for incongruent and congruent stimuli)
working memory (short-term memory) | The test was performed for each participant on day one and two at three predefined time points 9 a.m. (t1), 1 p.m. (t3), 5 p.m. (t5)
  Working memory was assessed with the Digit Span Backwards, in which participants are presented with a series of digits and then asked to recall them in reverse order. The main outcome for this test is the memory span.
sustained attention and vigilance | The test was performed for each participant on day one and two at three predefined time points 9 a.m. (t1), 1 p.m. (t3), 5 p.m. (t5)
  Sustained attention and vigilance were assessed with the Psychomotor Vigilance Task. Participants are presented with a visual stimulus (a simple light) that appears at random inter-stimulus intervals (between 2 and 10 seconds). When the stimulus appears, the participants are required to respond as quickly as possible. The primary outcome for this test is the mean reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, Study Director — University of Padua Department of Biomedical Sciences
Locations (1):
- Department of Biomedical Sciences, University of Padua, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No